CLINICAL TRIAL: NCT05712356
Title: A Phase 2a, Double-blind, Placebo-controlled, Multi-center, Randomized Study Evaluating LSTA1 When Added to Standard of Care (SoC) Versus Standard of Care Alone in Subjects With Advanced Solid Tumors (BOLSTER)
Brief Title: A Study of LSTA1 When Added to Standard of Care Versus Standard of Care Alone in Patients With Advanced Solid Tumors
Acronym: BOLSTER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LSTA1-P02; 2023-503740-14 (EudraCT Number)
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Cholangiocarcinoma; Gallbladder Cancer; Gallbladder Carcinoma; Intrahepatic Cholangiocarcinoma; Extrahepatic Cholangiocarcinoma; Bile Duct Cancer; Gall Bladder Cancer; Gall Bladder Carcinoma
Keywords: immunotherapy; chemo; chemotherapy; first line; second line; progression
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms; Bile Duct Neoplasms; Disease Progression | interventions — durvalumab; Cisplatin; Gemcitabine; Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LSTA1 arm for Untreated Cholangiocarcinoma (Experimental)
  Interventions: Drug: certepetide; Drug: Durvalumab; Drug: Cisplatin; Drug: Gemcitabine
- LSTA1 arm for Second-Line Cholangiocarcinoma (Experimental)
  Interventions: Drug: certepetide; Drug: FOLFOX regimen
- Placebo arm for Untreated Cholangiocarcinoma (Placebo Comparator)
  Interventions: Drug: Durvalumab; Drug: Cisplatin; Drug: Gemcitabine; Drug: Placebo
- Placebo arm for Second-Line Cholangiocarcinoma (Placebo Comparator)
  Interventions: Drug: FOLFOX regimen; Drug: Placebo

INTERVENTIONS:
Drug: certepetide — LSTA1 3.2 mg/kg given as a slow IV push over 1 minute when standard treatment(s) are given
  Other Names: CEND-1; LSTA1
  Arms: LSTA1 arm for Second-Line Cholangiocarcinoma; LSTA1 arm for Untreated Cholangiocarcinoma
Drug: Durvalumab — 1500 mg of durvalumab IV administered over 1 hour every 21 days for 8 cycles then every 28 days for additional cycles
  Other Names: Imfinzi
  Arms: LSTA1 arm for Untreated Cholangiocarcinoma; Placebo arm for Untreated Cholangiocarcinoma
Drug: Cisplatin — cisplatin 25 mg/m² IV administered over 30 minutes on day 1 and day 8 every 21 days for up to 8 cycles
  Arms: LSTA1 arm for Untreated Cholangiocarcinoma; Placebo arm for Untreated Cholangiocarcinoma
Drug: Gemcitabine — gemcitabine 1000 mg/m² IV administered over 30 minutes on day 1 and day 8 every 21 days for up to 8 cycles
  Arms: LSTA1 arm for Untreated Cholangiocarcinoma; Placebo arm for Untreated Cholangiocarcinoma
Drug: FOLFOX regimen — The following will be given every 14 days:
  * oxaliplatin 85 mg/m² and l-folinic acid 200 mg/m² or d,l-folinic acid 400 mg/m² concurrently, as a 2-hour IV infusion
  * fluorouracil (5-FU) 400 mg/m² will be given as an IV bolus over 5 minutes
  * fluorouracil (5-FU) 2400 mg/m² will be administered over 46 hours (via home-infusion pump)
  Other Names: Oxaliplatin; Folinic acid; Fluorouracil
  Arms: LSTA1 arm for Second-Line Cholangiocarcinoma; Placebo arm for Second-Line Cholangiocarcinoma
Drug: Placebo — Placebo given as a slow IV push over 1 minute when standard treatment(s) are given
  Arms: Placebo arm for Second-Line Cholangiocarcinoma; Placebo arm for Untreated Cholangiocarcinoma

SUMMARY:
The goal of this clinical trial is to test a new drug plus standard treatment compared with standard treatment alone in patients with previously untreated cholangiocarcinoma or those that have progressed after first-line treatment for cholangiocarcinoma.

The main questions it aims to answer are:

* is the new drug plus standard treatment safe and tolerable
* is the new drug plus standard treatment more effective than standard treatment

DETAILED DESCRIPTION:
This is a Phase 2a, double-blind, placebo-controlled, multi-center, randomized study of LSTA1 when added to standard of care (SoC) versus SoC alone in patients with advanced solid tumors. The study will include patients with previously untreated cholangiocarcinoma or those that have progressed after first-line treatment for cholangiocarcinoma.

The study will consist of a screening period, a run-in period, a treatment period, an end-of-treatment follow-up visit, and a long-term follow up period.

Participants who provide informed consent will be screened for eligibility within 28 days prior to beginning the study treatment run-in period. Once eligibility is confirmed, participants will be randomized to one of the two treatment groups (SoC + placebo vs. SoC + LSTA1).

During the 3-day run-in period, participants will only receive the LSTA1 or placebo components of their randomized treatment regimen. After the 3-day run-in, Cycle 1 of treatment will commence. Tumor scans will be performed every 8 weeks (56 days ± 7 days) while on treatment.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy ≥ 3 months
* At least one measurable lesion as assessed by RECIST 1.1
* Adequate organ and marrow function
* Adequate contraception
* Patients with either of the following:

  * Pathologically confirmed metastatic or unresectable cholangiocarcinoma or gallbladder carcinoma (GBC), with no prior systemic chemotherapy or targeted therapy or loco-regional therapy (including but not limited to transarterial chemoembolization, transarterial embolization, transarterial chemotherapy or transarterial radioembolization). Patients with recurrent disease more than 6 months after completion of adjuvant chemotherapy following curative resection are eligible.
  * Pathologically confirmed metastatic or unresectable cholangiocarcinoma or GBC with progression of disease after first-line chemotherapy and immunotherapy.

Exclusion Criteria:

* Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results, including but not limited to:

  * Any major surgery or irradiation less than 4 weeks prior to baseline disease assessment
  * Active infection (viral, fungal, or bacterial) requiring systemic therapy
  * Known active hepatitis B virus, hepatitis C virus, or HIV infection
  * Active tuberculosis as defined per local guidance
  * History of allogeneic tissue/solid organ transplant
  * Prior malignancy requiring active treatment within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
  * Pregnant or breastfeeding
  * Clinically significant or symptomatic cardiovascular/cerebrovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) within 6 months before randomization
* History or clinical evidence of symptomatic central nervous system (CNS) metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 30 days after treatment discontinuation
  The National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE) will be used to grade the intensity of adverse events throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Kristen K Buck, MD, Study Chair — Lisata Therapeutics, Inc.
Locations (19):
- United States (19):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Moffitt Cancer Center, Tampa, Florida
  - Alliance for Multispecialty Research, Merriam, Kansas
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - Norton Cancer Institute, Audubon, Louisville, Kentucky
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Northwell Health - Zuckerberg Cancer Center, Lake Success, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - FirstHealth of the Carolinas, Inc., Pinehurst, North Carolina
  - Carl & Edyth Lindner Center for Research & Education at The Christ Hospital and The Christ Hospital Cancer Center, Cincinnati, Ohio
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia